CLINICAL TRIAL: NCT03638323
Title: Pilot Study of the Links Between Presbyacusis and Lexical Disorders in Patients With Alzheimer's Disease or Related Disease
Brief Title: Age-related Hearing Loss and Lexical Disorders
Acronym: LOOP
Status: Completed | Type: Observational
Sponsor: Groupe Hospitalier de la Rochelle Ré Aunis (Other)
Responsible Party: Sponsor
Other Study IDs: 2018/P08/256
Record Dates: First submitted 2018-08-14; First posted 2018-08-20 (Actual); Results first posted 2019-09-11 (Actual); Last update posted 2019-12-05 (Actual); Status verified 2019-11

CONDITIONS: Alzheimer Disease; Presbycusis; Lexical Syntactic Disorder
MeSH Terms: conditions — Alzheimer Disease; Presbycusis | interventions — Speech Therapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LOOP group: Speech therapy consultation for patients with Alzheimer's disease
  Interventions: Other: Speech therapy

INTERVENTIONS:
Other: Speech therapy — During a 1-hour speech-language consultation, a lack of word evaluation will be conducted and patient will answer a Hearing Difficulty Questionnaire

SUMMARY:
In France, Alzheimer's disease accounts for 70 to 80% of the causes of neurocognitive disorders, i.e. 600,000 to 800,000 patients. It is a neurodegenerative pathology that causes evolutionary cognitive dysfunction, mainly affecting memory functions. The inability to name familiar objects (lack of the word) is one of the most commonly noted symptoms at an early stage of the disease.

Presbyacusis, or age-related hearing loss, is the most common sensory deficit in the elderly which is manifested socially by a progressive discomfort of verbal communication. Presbyacusis remains underdiagnosed and undertreated: 2/3 of the patients are not using hearing aid.

In recent years, a link between neurocognitive disorders and hearing loss has been shown by investigating general cognition. In this study, the investigators are investigating lexical disorders.

ELIGIBILITY:
Inclusion Criteria:

* > 65 years old
* French mother tongue
* Good vision with or without correction
* Alzheimer's or related disease (15 <Mini-Mental State Examination<25)
* Affiliate or beneficiary of a social security
* Informed consent

Exclusion Criteria:

* Cognitive disorders related to another pathology (cerebrovascular accident, head trauma, epilepsy ...)
* Protected patient (under guardianship) or person deprived of liberty by judicial or administrative decision

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Series of patients from the Care Center for the Elderly (geriatric day hospital, long-term care units, follow-up care units and rehabilitation)
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2018-08-27 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Laure Vignaud, Ph.D., Study Director — Groupe Hospitalier de la Rochelle Ré Aunis
Locations (1):
- Groupe Hospitalier de la Rochelle Ré Aunis, La Rochelle, France

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Number of screend patients: 46 Number of patient excluded: 9
  * 1 refusal
  * 7 lack an inclusion criteria or had an exclusion criteria
  * 1 was excluded after enrolment due to comprehension disorders and unreliable responses to the Hearing Questionnaire
Period: Overall Study
Arm/Group | LOOP Group
Started | 38
Completed | 37
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- Normal Hearing: Participants were divided into two groups based on their score on the Hearing Questionnaire. Patients with a score of less than 14 are in the "normal hearing" group
- Risk of Presbycusis: Participants were divided into two groups based on their score on the Hearing Questionnaire. Patients with a score of 14 or more are in the "risk of presbycusis" group
- Total: Total of all reporting groups
Arm/Group | Normal Hearing | Risk of Presbycusis | Total
Number analyzed (Participants) | 29 | 8 | 37
Age, Continuous [Median (Full Range); unit: years] | 78 [68 to 87] | 80.5 [71 to 86] | 79 [68 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 6 | 25
  Male | 10 | 2 | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Educational level [Count of Participants; unit: Participants]
  Certificate study | 18 | 5 | 23
  baccalaureat or more | 11 | 3 | 14
Residency [Count of Participants; unit: Participants]
  At home | 29 | 7 | 36
  Institution | 0 | 1 | 1
Laterality [Count of Participants; unit: Participants]
  left handed | 3 | 0 | 3
  right handed | 26 | 8 | 34
Diagnostic [Count of Participants; unit: Participants]
  Alzheimer's disease | 7 | 3 | 10
  Related disease | 22 | 5 | 27
Hearing aid [Count of Participants; unit: Participants]
  yes | 1 | 2 | 3
  no | 28 | 6 | 34
Speech and language therapy [Count of Participants; unit: Participants]
  yes | 6 | 4 | 10
  no | 23 | 4 | 27

OUTCOME MEASURES:

1. Primary Outcome: Link Between Lack of Word and Presbycusis
Description: The Batterie Informatisée du Manque du Mot (BIMM) is a computerized assessment instrument for denominational disorders. It provides information on level of lexical impairment, type of error (phonological, semantic, visual perceptual) and response time. It comprises two tests: denomination of nouns (42 items, score range from 0 to 42) and of verbs (28 items, score range from 0 to 28). The results are presented in a report including scores, description of qualitative errors, and results per item. A global score of less than 40 indicates a lack of words. The score range is between 0 and 70.
  The hearing questionnaire consists in 14 questions about concrete situations and a direct question about what the patient thinks of his hearing. Answers are quoted 0, 2 or 4 points. An overall score greater than 14 indicates presbycusis.
Time Frame: at inclusion
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Normal Hearing | Risk of Presbycusis
Number analyzed (Participants) | 29 | 8
score on a scale
  Global score | 38 [21 to 50] | 38.5 [24 to 50]
  Score at denomination of nouns | 23 [12 to 30] | 21.5 [15 to 32]
  Score at denomination of verbs | 15 [9 to 20] | 17 [9 to 19]

2. Secondary Outcome: Association Between Age and Lack of Word
Description: Age of patients and score at the lack of word questionnaire (BIMM) The Batterie Informatisée du Manque du Mot (BIMM) is a computerized assessment instrument for denominational disorders. It provides information on level of lexical impairment, type of error (phonological, semantic, visual perceptual) and response time. It comprises two tests: denomination of nouns (42 items) and of verbs (28 items). The results are presented in a report including scores, description of qualitative errors, and results per item. An score less than 40 indicates lack of word.
Time Frame: at inclusion
Measure: Median (Full Range); unit: years
Groups:
- No Word Alteration: Patients with a score of 40 or more at the BIMM questionnaire are in the "no word alteration" group
- Lack of Word: Patients with a score of less than 40 at the BIMM questionnaire are in the "lack of word" group
Arm/Group | No Word Alteration | Lack of Word
Number analyzed (Participants) | 19 | 24
years | 76 [68 to 87] | 80 [72 to 86]

3. Secondary Outcome: Association Between Gender and Lack of Word
Description: Male or female and score at the lack of word questionnaire (BIMM) The Batterie Informatisée du Manque du Mot (BIMM) is a computerized assessment instrument for denominational disorders. It provides information on level of lexical impairment, type of error (phonological, semantic, visual perceptual) and response time. It comprises two tests: denomination of nouns (42 items) and of verbs (28 items). The results are presented in a report including scores, description of qualitative errors, and results per item. An score less than 40 indicates lack of word.
Time Frame: at inclusion
Measure: Count of Participants; unit: Participants
Arm/Group | No Word Alteration | Lack of Word
Number analyzed (Participants) | 16 | 21
Participants
  Female | 7 | 18
  Male | 9 | 3

4. Secondary Outcome: Association Between Study Level and Lack of Word
Description: Primary (certificate study), secondary and tertiary study (baccalaureat and more) level and score at the lack of word questionnaire (BIMM) The Batterie Informatisée du Manque du Mot (BIMM) is a computerized assessment instrument for denominational disorders. It provides information on level of lexical impairment, type of error (phonological, semantic, visual perceptual) and response time. It comprises two tests: denomination of nouns (42 items) and of verbs (28 items). The results are presented in a report including scores, description of qualitative errors, and results per item. An score less than 40 indicates lack of word.
Time Frame: at inclusion
Measure: Count of Participants; unit: Participants
Arm/Group | No Word Alteration | Lack of Word
Number analyzed (Participants) | 16 | 21
Participants
  Primary level | 6 | 17
  Secondary & tertiary level | 10 | 4

5. Secondary Outcome: Association Between Accommodation Type and Lack of Word
Description: Patient living at home or in an institution and score at the lack of word questionnaire (BIMM) The Batterie Informatisée du Manque du Mot (BIMM) is a computerized assessment instrument for denominational disorders. It provides information on level of lexical impairment, type of error (phonological, semantic, visual perceptual) and response time. It comprises two tests: denomination of nouns (42 items) and of verbs (28 items). The results are presented in a report including scores, description of qualitative errors, and results per item. An score less than 40 indicates lack of word.
Time Frame: at inclusion
Measure: Count of Participants; unit: Participants
Arm/Group | No Word Alteration | Lack of Word
Number analyzed (Participants) | 16 | 21
Participants
  At home | 15 | 21
  Institution | 1 | 0

6. Secondary Outcome: Association Between Laterality and Lack of Word
Description: Right or left handed patients and score at the lack of word questionnaire (BIMM) The Batterie Informatisée du Manque du Mot (BIMM) is a computerized assessment instrument for denominational disorders. It provides information on level of lexical impairment, type of error (phonological, semantic, visual perceptual) and response time. It comprises two tests: denomination of nouns (42 items) and of verbs (28 items). The results are presented in a report including scores, description of qualitative errors, and results per item. An score less than 40 indicates lack of word.
Time Frame: at inclusion
Measure: Count of Participants; unit: Participants
Arm/Group | No Word Alteration | Lack of Word
Number analyzed (Participants) | 16 | 21
Participants
  Right handed | 16 | 18
  Left handed | 0 | 3

7. Secondary Outcome: Association Between Main Diagnosis and Lack of Word
Description: Alzheimer's disease or related disease and score at the lack of word questionnaire (BIMM) The Batterie Informatisée du Manque du Mot (BIMM) is a computerized assessment instrument for denominational disorders. It provides information on level of lexical impairment, type of error (phonological, semantic, visual perceptual) and response time. It comprises two tests: denomination of nouns (42 items) and of verbs (28 items). The results are presented in a report including scores, description of qualitative errors, and results per item. An score less than 40 indicates lack of word.
Time Frame: at inclusion
Measure: Count of Participants; unit: Participants
Arm/Group | No Word Alteration | Lack of Word
Number analyzed (Participants) | 16 | 21
Participants
  Alzheimer's disease | 3 | 7
  Related disease | 13 | 14

8. Secondary Outcome: Association Between Hearing Aid and Lack of Word
Description: Patients with or without hearing aid and score at the lack of word questionnaire (BIMM) The Batterie Informatisée du Manque du Mot (BIMM) is a computerized assessment instrument for denominational disorders. It provides information on level of lexical impairment, type of error (phonological, semantic, visual perceptual) and response time. It comprises two tests: denomination of nouns (42 items) and of verbs (28 items). The results are presented in a report including scores, description of qualitative errors, and results per item. An score less than 40 indicates lack of word.
Time Frame: at inclusion
Measure: Count of Participants; unit: Participants
Arm/Group | No Word Alteration | Lack of Word
Number analyzed (Participants) | 16 | 21
Participants
  yes | 0 | 3
  no | 16 | 18

9. Secondary Outcome: Association Between Speech Therapy and Lack of Word
Description: Patients with or without ongoing speech therapy and score at the lack of word questionnaire (BIMM) The Batterie Informatisée du Manque du Mot (BIMM) is a computerized assessment instrument for denominational disorders. It provides information on level of lexical impairment, type of error (phonological, semantic, visual perceptual) and response time. It comprises two tests: denomination of nouns (42 items) and of verbs (28 items). The results are presented in a report including scores, description of qualitative errors, and results per item. An score less than 40 indicates lack of word.
Time Frame: at inclusion
Measure: Count of Participants; unit: Participants
Arm/Group | No Word Alteration | Lack of Word
Number analyzed (Participants) | 16 | 21
Participants
  yes | 5 | 5
  no | 11 | 16

ADVERSE EVENTS:
Time Frame: 5 months
Arm/Group | LOOP Group
All-Cause Mortality (participants affected / at risk) | 0/37
Serious Adverse Events (participants affected / at risk) | 0/37
Other Adverse Events (participants affected / at risk) | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-08): https://cdn.clinicaltrials.gov/large-docs/23/NCT03638323/Prot_SAP_000.pdf